CLINICAL TRIAL: NCT05382507
Title: The Ultrasonographic Measurement of Quadriceps Muscle Thickness and the Shape of the Femoral Nerve in Patients Undergoing Total Knee Arthroplasty: an Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0229
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For each individual, the femoral nerve shows various shapes and locations. This is because the femoral nerve is located on top of the iliacus muscle, so the shape and location of the femoral nerve seems to be related to the patient's muscle mass. Ultrasound of the quadriceps femoris could represent a widely available, non-invasive, affordable, and reliable tool to evaluate skeletal muscle. We aim to investigate the relationship between muscle mass and the shape of the femoral nerve through this observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years old or older and scheduled for elective total knee arthroplasty

Exclusion Criteria:

1. Pre-existing neurologic or anatomic deficits in the lower extremities

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
the thickness of rectus femoralis and vastus intermedius, the shape of the femoral nerve | preoperative (about 10 minutes before entering the operating room)
  Assessment of quadriceps femoris thickness using ultrasound. Thickness of each muscle is measured from the femur to the inner edge of the vastus intermedius (VI) muscle, or from subcutaneous tissue to the inner edge of the rectus femoris (RF) muscle. The shape of the femoral nerve was measured by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Bora Lee, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No